CLINICAL TRIAL: NCT05954000
Title: Reducing African-American CVD Disparities Intervention Optimization (RADIO) Program: A Dose Finding Pilot Study Protocol and Focus Group Results
Brief Title: Reducing African-American CVD Disparities Intervention Optimization (RADIO) Individuals on Statins
Acronym: RADIO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Toronto Dominion Bank (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 21-1192
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Medication Adherence
Keywords: medication; adherence; dose finding; personalized; digital; TiTE-CRM
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: The study utilizes a modified Time-To-Event Continual Reassessment Method Dose-Finding Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Dose-finding study with 14 groups of 3 participants each. To identify the minimum effective dose (MED) to increase medication adherence by 20% between run-in and follow-up periods, the first group of 3 participants will receive a 5-week dose of the multi-BCT intervention. For the next subjects, the doses to administrate will vary between 1 and 10 weeks in length and will be determined by the modified Time-to-Event Continual Reassessment Method (TiTE-CRM) according to the observed responses in the previous subjects.
  Interventions: Behavioral: 5 Behavioral Change Techniques

INTERVENTIONS:
Behavioral: 5 Behavioral Change Techniques — 1. Goal setting: set or agree on a goal defined in terms of behavior to be achieved. Example: Set the goal to take your medication as prescribed tomorrow.
  2. Action planning: prompt detailed planning of performance of behavior (must include a setting, frequency, duration, and intensity). Example: Develop a plan for taking your medication.
  3. Self-Monitoring of behavior: establish a method for person to monitor and record their behavior. Example: Did you take your statin medication today?
  4. Feedback on behavior: Monitor and provide informative or evaluative feedback on performance of the behavior (e.g. form, frequency, duration, intensity). Example: You did not take your statin medication as prescribed yesterday.
  5. Prompts/Cues: introduce or define environmental or social stimulus with the purpose of prompting or cueing the behavior. The prompt or cue would normally occur at the time or place of performance. Example: Please remember to take your medication soon.

SUMMARY:
The purpose of this project is to identify the minimum effective dose (MED) of a multi-component behavioral change intervention required to increase levels of medication adherence among Black and African American individuals on primary prevention statin therapy who are at elevated risk for cardiovascular disease (CVD). The intervention will be comprised of 5 BCTs which have previously shown to be effective on increasing health behaviors: Goal Setting, Action Planning, Self-Monitoring, Feedback, and Prompts/Cues. Participants will complete a 2-week run-in period where medication adherence levels will be measured using a smart pill bottle and physical activity (PA) will be measured using Fitbit wearable devices. Then 42 participants will be randomized into 14 cohorts of 3 participants each for the intervention period. During the intervention period, participants will receive a multi-BCT intervention, the length of which varies between 1 and 10 weeks depending on the assigned dose. Assignment to doses will utilize a modified version of the Time-to-Event Continual Reassessment Method (TiTE-CRM) methodology to adjust the dose for each cohort based on the results from the previous cohort. After the intervention, there will be a 2-week follow-up period. The MED will be defined as the smallest BCT dose (defined by weeks of intervention) associated with 80% of participants having a 20% medication adherence increase between the run-in and the follow-up periods. The long-term goal is reduce incidence of CVD among Black and African American individuals by increasing adherence to primary prevention statin medications.

DETAILED DESCRIPTION:
The purpose of this project is to identify the minimum effective dose (MED) of a multi-component behavioral change technique (BCT) intervention required to increase statin medication adherence among Black and African American individuals on primary prevention statin therapy who are at elevated risk for cardiovascular disease (CVD). The long-term goal is to prevent CVD among Black and African American individuals. The current project will utilize a modified version of the time-to-event continual reassessment method (TiTE-CRM), a state of the art dose finding methodology, to determine the MED of a multi-component BCT intervention required to increase the proportion of days adherent to statin medications by 20%. The intervention will be comprised of 5 BCTs which have previously shown to be effective on increasing health behaviors: Goal Setting, Action Planning, Self-Monitoring, Feedback, and Prompts/Cues.

The study sample will include individuals who identify as Black or African American and are currently prescribed primary prevention statin therapy. For this research, the investigators will enroll participants with low levels of self-reported adherence to statin medications, with the goal of randomizing 42 persons to the intervention. Enrolled participants will complete a 2-week run-in period where levels of adherence to statin medications will be assessed using a smart pill bottle and physical activity levels will be measured using a Fitbit wearable device. During the run-in period, data from the smart pill bottle will be used to verify objective non-adherence to statin medications (defined as taking statin medications as prescribed for less than 80% of days). Individuals who do not meet objective levels of nonadherence to statin medications and/or are non-adherent to the protocol will be excluded and will not be randomized to the intervention. Following the run-in, the investigators will randomize 42 participants into 14 cohorts of 3 participants each for the intervention period. During the intervention period, participants will receive a multi-BCT intervention, the length of which varies between 1 and 10 weeks depending on the assigned dose of a multi-BCT intervention. Assignment to doses will utilize modified TiTE-CRM methodology to adjust the dose for each cohort based on the results from the previous cohort. Following the intervention, all participants will be assessed over a 2-week follow-up period which includes passive data collection from the activity monitor, answering surveys and use of the electronic pill bottle to track medication adherence. The MED will be defined as the smallest BCT dose duration associated with a 20% increase in the proportion of days using statin medication as prescribed between the run-in and the follow-up periods in 80% of the sample receiving that dose. Adherence to statins will be defined using changes in weight of medication in the smart pill bottle. The investigators will also assess Mechanisms of Action (MoAs) to determine potential mediators of the BCT intervention on physical activity (PA). As some evidence suggests there are correlations between adherence and PA and that interventions targeting medication adherence also influence PA, the investigators will utilize Fitbit devices to determine whether the BCT intervention increase participant's levels of activity.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as Black/African American
* Aged ≥ 18 years
* Speaks English
* Has a self-report of low adherence to statin medication
* Prescribed statin medication
* Owns and can regularly access a smartphone capable of receiving text messages and accessing the internet
* Ambulatory without limitations (has never been advised by a clinician that increasing low-intensity walking would be unsafe)

Exclusion Criteria:

* History of CVD
* Does not speak English
* Does not own or cannot regularly access a smartphone capable of receiving text messages
* Inability to comply with study protocol during a 2-week run-in period
* Unavailable for follow-up
* Cognitive impairment; severe mental illness (e.g., bipolar disorder or schizophrenia)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Success or failure for change in Medication Adherence. | Medication adherence will be assessed continuously via the smart pill bottle and adherence will be calculated daily. The change in proportion of days adherent will be compared between the run-in and follow-up periods (5-14 weeks from run-in).
  Participant medication adherence increase will be assessed between run-in and follow-up periods using the smart pill bottle. A successful adherence increase is defined as average daily adherence to statin medications in the 2-week follow-up period being higher by 20% or more than in the 2-week run-in period. The minimum effective dose (MED) will be defined as the smallest BCT dose duration associated with 80% of participants receiving that dose having a successful statin adherence increase between the run-in and the follow-up periods.

SECONDARY OUTCOMES:
Within-person change in Medication Adherence. | Medication adherence will be assessed continuously via a smart pill bottle and adherence will be calculated daily. Change over time will be examined between the baseline, intervention, and follow-up periods (5-14 weeks from run-in).
  Participant adherence to stain medication will be assessed continuously using a smart electronic pill bottle. Daily medication adherence will be recorded for each participant across the full duration of the study. Changes in medication between run-in and intervention phases will be compared using Generalized Linear Mixed Model Analyses.
Within-person change in Self-Efficacy. | Self-efficacy will be assessed at the completion of baseline and will be assessed every 2 weeks until the end of the follow-up period (5-14 weeks from run-in).
  Self-efficacy will be assessed using an adapted version of the PROMIS Item Bank v1.0, Self-Efficacy for Managing Chronic Conditions, Managing Medications and Treatment Short Form 8a, a 7-item measure assessing patient's capabilities to take their medications. Items are scored on a 1 "I am not at all confident" to 5 "I am very confident" scale. Scale scores will be converted to T-scores using methods from the PROMIS scoring manual based on item response theory, with higher scores indicating higher levels of self-efficacy.
Within-person change in Behavioral Automaticity. | Behavioral automaticity will be assessed at the completion of baseline and will be assessed every 2 weeks until the end of the follow-up period (5-14 weeks from run-in)
  Behavioral automaticity will be assessed using an adapted version of the 4-item Self-Report Behavioral Automaticity Index (SRBAI) which assesses automaticity of behavior. Items are scored on a 1 "Strongly Disagree" to 7 "Strongly agree" scale, and summed to create a total score, with higher scores indicating greater behavioral automaticity.
Within-person change in Discrepancy in Behavior. | Feedback Processes will be assessed at the completion of baseline and will be assessed every 2 weeks until the end of the follow-up period (5-14 weeks from run-in).
  This will be assessed with a single item stating "How large is the difference between your current medication taking behavior and the frequency of medication use prescribed by your doctor?" This item is rated on a scale of 1 "Not at all different" to 7 "Very different", with higher scores indicating greater levels of discrepancy in behavior.
Within-person change in Environmental Context and Resources. | Environmental Context and Resources will be assessed at the completion of baseline and will be assessed every 2 weeks until the end of the follow-up period (5-14 weeks from run-in).
  Environmental context and resources will be assessed using a list of 4 potential environmental barriers to medication adherence taken from Fung and colleagues. Barriers are rated on a 1 "Not often at all" to 5 (Very often) scale, and summed to create a total score, with higher scores indicating that the listed barriers had greater effects on patient nonadherence to statins.
Within-person change in Motivation. | Motivation will be assessed at the completion of baseline and will be assessed every 2 weeks until the end of the follow-up period (5-14 weeks from run-in).
  Motivation will be assessed with a message stating "I feel motivated to take my statin medications exactly as my doctor prescribed." Motivation will be rated on a scale of 1 "Not at all true" to 7 "Very True", with higher scores indicating greater levels of motivation.
Within-person change in Daily Steps. | Steps will be assessed continuously via worn activity tracker and step counts will be calculated daily. Change over time will be examined between the baseline, intervention, and follow-up periods (5-14 weeks from run-in)
  Participant steps will be assessed continuously using a Fitbit mobile device. Daily steps for participants will be aggregated by run-in and follow-up periods to generate average daily steps in each period. Changes in daily steps between run-in and intervention periods will be compared using Generalized Linear Mixed Model Analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Butler, PhD, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD) will be de-identified and pooled before sharing on the Open Science Framework, along with a data dictionary. Pooling trials together is a more efficient approach for deriving population-level estimates than conventional randomized controlled trials.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol, including the statistical analysis plan, will be made available in addition to the informed consent form following completion of recruitment but prior to publication of any data from the current study. De-identified, pooled individual participant data will be made available within a year of final participant data collection. We anticipate this data to be available on the Open Science Framework platform indefinitely.
Access Criteria: All data and supporting information will be stored on the Open Science Framework, a free web application with no access restrictions.

DOCUMENTS (1):
  • Informed Consent Form (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT05954000/ICF_000.pdf